CLINICAL TRIAL: NCT03507101
Title: Invasive Disease Caused by Group A Streptococcus (GAS) - a Prospective Study (DICAR)
Brief Title: Invasive Disease Caused by Group A Streptococcus (GAS) (DICAR)
Acronym: DICAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); University of Turku (Other)
Responsible Party: Principal Investigator, Ville Kaila, Clinical investigator, Tampere University Hospital
Other Study IDs: DICAR
Record Dates: First submitted 2018-04-19; First posted 2018-04-24 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Invasive Group A Beta-Haemolytic Streptococcal Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will obtain DNA and RNA samples from all study patients for genetic and transcriptomic analysis to assess inherited risk factors and immunologic response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasive GAS infection study patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No particular intervention or exposure is of particular interest

SUMMARY:
The goal of this study is to gain important knowledge on the pathogenesis and prognostic factors in severe invasive group A streptococcal (GAS) infections, as well as the effects of individual characteristics of both the pathogen and the patient on disease severity. The aim is to recruit a minimum of 60 patients from Tampere and Turku University Hospitals in 2-3 years to gather a suitably wide spectrum of manifestations of the disease, and gather genetic, transcriptomic and diagnostic data on both the patients and pathogens in an effort to further our understanding of the pathogenesis of severe invasive GAS disease.

DETAILED DESCRIPTION:
Invasive group A streptococcal (GAS) infection is a severe, life threatening disease. New prognostic markers are needed to better identify patients at risk of severe complications to better improve their care. By advancing understanding of the mechanisms of severe disease, treatments may be found to hinder the processes behind them. It is likely that different individuals react differently to the same microbe.

From previous incidence data the investigators have estimated that it will be possible to recruit a minimum of 60 patients over the course of 2-3 years from Tampere and Turku University Hospitals. This sample size should contain a reasonably wide array of infections with varying stages of severity. The investigators will then gather genetic and transcriptomic data on these patients at three time points, as well as salival samples for antibody analysis, and throat cultures to screen for carriage of the pathogen in question. The genome of all the GAS strains obtained from the patients will also be sequenced. From this the investigators hope to derive information pertaining to the interplay of the patients immunologic response and the pathogens inherent characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have been diagnosed with invasive group A streptococcal disease and are willing to participate

Exclusion Criteria:

* Underage patients are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 60 patients from Tampere and Turku University Hospitals who contract invasive group A streptococcal disease within our recruitment period. The size of the study population has been difficult to calculate exactly, but the investigators have gauged the size according to previous epidemiological data to have a population that has a wide variety of disease courses to get a good understanding of the pathogenesis, and that can be recruited within 2-3 years.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Severe invasive GAS disease | Four month follow up
  GAS infection leading to death, complications or disability

CONTACTS AND LOCATIONS:
Overall Officials: Jaana Syrjänen, PhD, Study Director — Tampere University Hospital
Locations (2):
- Finland (2):
  - Tampere university hospital, Tampere, Pirkanmaa
  - Turku university hospital, Turku, Southwest Finland

IPD SHARING:
Plan to Share IPD: Undecided
In the future it may be possible to make this data available to continue research under this topic. In such a case a request would have to be made through the review board of the Tampere University Hospital.

REFERENCES:
- [Derived] Kailankangas V, Vilhonen J, Grondahl-Yli-Hannuksela K, Rantakokko-Jalava K, Seiskari T, Auranen K, Lonnqvist E, Virolainen M, Hyyrylainen HL, Oksi J, Syrjanen J, Vuopio J. Presence of Streptococcus pyogenes in the throat in invasive Group A Streptococcal disease: a prospective two-year study in two health districts, Finland. Infect Dis (Lond). 2023 Jun;55(6):405-414. doi: 10.1080/23744235.2023.2192287. Epub 2023 Apr 8. PMID 37029930